CLINICAL TRIAL: NCT04144374
Title: Comparison of Omadacycline Pharmacokinetics and Soft-Tissue Penetration in Diabetic Patients With Wound Infections Versus Healthy Volunteers Via In Vivo Microdialysis
Brief Title: Omadacycline Tissue Penetration in Diabetic Patients With Wound Infections and Healthy Volunteers Via In Vivo Microdialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HHC-2019-0220
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Diabetes; Wound Infection; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus; Wound Infection | interventions — omadacycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetic Wound Infection (Experimental): Participants with a documented medical history of Type 1 or Type 2 diabetes and a mild to moderate (Grade 2 or 3) wound infection of the lower limb will receive 3 to 5 doses of omadacycline once daily, followed by sampling of interstitial tissue fluid at the margin of the wound by a microdialysis probe over 24 hours following the last dose (e.g., 48-72 hours).
  Interventions: Drug: Omadacycline; Procedure: Microdialysis Catheter Insertion
- Healthy Volunteers (Active Comparator): Participants will be male or female healthy adult volunteers with no significant medical or medication history. Participants will receive 3 doses of omadacycline once daily, followed by sampling of interstitial tissue fluid at the margin of the wound by a microdialysis probe over 24 hours following the last dose (e.g., 48-72 hours).
  Interventions: Drug: Omadacycline; Procedure: Microdialysis Catheter Insertion

INTERVENTIONS:
Drug: Omadacycline — Omadacycline will be administered 200 mg IV once daily on day 1 followed by omadacycline 300 mg by mouth once daily for 2-4 doses.
  Other Names: Nuzyra
Procedure: Microdialysis Catheter Insertion — A 20 kilodalton microdialysis probe (63 MD catheter; MDialysis Inc., N. Chelmsford, MA) will be inserted into the subcutaneous tissue at the margin of the wound (patient group) or in the thigh tissue (healthy volunteers). The probe will be left in place for the final dose and all tissue sampling procedures thereafter. This probe is perfused with a physiologic solution to collect interstitial fluid samples. The probe will then be removed after completion of sample collection.

SUMMARY:
This study will determine the tissue penetration of the novel tetracycline antibiotic, omadacycline (Nuzyra, Paratek Pharmaceuticals, Inc.), into the extracellular, interstitial fluid of soft tissue in diabetic patients with lower limb wound infections. Penetration will be compared with a group of healthy volunteer control participants.

DETAILED DESCRIPTION:
This study will enroll 10 patients with diabetes who are admitted with a lower limb wound infection and 6 healthy volunteer control participants. The study will take place in an inpatient unit at Hartford Hospital for all patients and in the Clinical Research Center at Hartford Hospital for all healthy volunteers. All participants will receive 3 to 5 doses of omadacycline (200mg IV once daily on day 1, transitioned to 300 mg by mouth thereafter). A microdialysis probe (Mdialysis Inc., N. Chelmsford, MA) will be inserted into the subcutaneous soft tissue near the margin of the wound (patients) or in the thigh (healthy volunteers). The microdialysis probe is perfused with normal saline solution and samples are collected for the 24 hours following the final dose (i.e., 48-72 hours). A peripheral intravenous catheter will be inserted into an arm vein to collect blood samples simultaneously with microdialysis samples. Concentrations in tissue are compared with blood to determine percent penetration.

ELIGIBILITY:
Inclusion Criteria:

Experimental: Type 1 or Type 2 diabetes and a mild to moderate (Grade 2 or 3) wound infection of the lower limb

Active Comparator: Healthy Adult Volunteer

Exclusion Criteria:

Participants in the study or control group will be excluded if any of the following criteria are met:

* Less than 18 years of age
* History of hypersensitivity to omadacycline or any tetracycline based molecule
* History of hypersensitivity to lidocaine or lidocaine derivatives
* Pregnant or breastfeeding
* Concomitant receipt of any tetracycline based antibiotic therapy
* Any other documented reason felt by the investigator to potentially affect the outcomes of the study

Additional Exclusion Criteria for Diabetic Patient Study Group:

* Participants likely to require multiple surgical interventions during the study period, which therefore could affect placement of the microdialysis catheter

Additional Criteria for Healthy Volunteer Control Group:

* Body Mass Index (BMI) ≥ 35 kg/m2
* Serum creatinine greater than 1.5 mg/dl or creatinine clearance (CrCl) < 50ml/min, as calculated by Cockroft-Gault using ideal body weight for all participants
* Presence of anemia, thrombocytopenia, or leukopenia as defined by hematocrit, platelet, or white blood cell count < 75% of the lower limit of normal
* Aspartate transaminase, alanine aminotransferase, or alkaline phosphatase greater than five times upper limit of normal
* Total bilirubin greater than three times the upper limit of normal
* Any known active co-morbidity listed on medical history or that becomes apparent during physical examination
* Positive urine drug screen (cocaine, THC, opiates, benzodiazepines, and amphetamines)
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
* Use of tobacco- or nicotine-containing products in excess of the equivalence of 5 cigarettes per day.
* Consumption of caffeine between Study Days 1 and 4
* Use of prescription or nonprescription drugs, vitamins, or dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, with the exception of acetaminophen at doses of ≤ 1 g/day. The use of hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Omadacycline Tissue Penetration. | 48-72 hours
  The ratio of omadacycline tissue concentrations to blood concentrations following the final omadacycline dose.

SECONDARY OUTCOMES:
Omadacycline Area Under the Curve (AUC) in Tissue | 48-72 hours
  he area under the drug concentration-time curve (AUC) in tissue reflects the actual tissue exposure to drug after administration of a dose of the drug and is expressed in mg*h/L. Venous blood was obtained via peripheral intravenous catheter at 48 hours from the start of the first dose (i.e., immediately before administration of the 3rd dose), and at 49, 50, 50.5, 51, 51.5, 52, 54, 56, 60, 64 and 72 hours. Dialysate samples of 120μL were collected in 200µL microvials simultaneously with plasma at 48, 49, 50, 51, 52, 53, 54, 55, 56, 57, 58, 59, 60, 64, 68 and 72 hours following administration of the first dose.

CONTACTS AND LOCATIONS:
Overall Officials: David P Nicolau, PharmD, Principal Investigator — Center for Anti-Infective Research and Development, Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No